CLINICAL TRIAL: NCT06020170
Title: Delving Into Participation Patterns in Social Anxiety Clinical Trials and Investigating Engagement Trends Among Individuals Impacted by the Disease
Brief Title: Delving Into Participation Patterns in Social Anxiety Studies
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 83342231
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Social Anxiety
Keywords: social anxiety

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study seeks to delve into the firsthand experiences of patients diagnosed with social anxiety who partake in a separate clinical trial featuring a specific medical intervention. The primary emphasis will be on meticulously tracking the rates of trial completion and withdrawal among these individuals.

By joining this clinical trial, individuals have the unique opportunity to contribute to the betterment of future social anxiety patients and play an active role in advancing medical research.

ELIGIBILITY:
Inclusion Criteria:

* Patient has self-identified as planning to enroll in a clinical trial
* Patient has been diagnosed with social anxiety
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Inability to perform regular electronic reporting
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with social anxiety who are actively considering enrolling in an observational clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in a social anxiety clinical trial | 3 months
Rate of patients who remain in social anxiety clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alvi T, Kumar D, Tabak BA. Social anxiety and behavioral assessments of social cognition: A systematic review. J Affect Disord. 2022 Aug 15;311:17-30. doi: 10.1016/j.jad.2022.04.130. Epub 2022 Apr 28. PMID 35490878
- [Background] Gao J, Feng Y, Xu S, Wilson A, Li H, Wang X, Sun X, Wang Y. Appearance anxiety and social anxiety: A mediated model of self-compassion. Front Public Health. 2023 Mar 21;11:1105428. doi: 10.3389/fpubh.2023.1105428. eCollection 2023. PMID 37026142
- [Background] Fancourt D, Steptoe A, Bu F. Trajectories of anxiety and depressive symptoms during enforced isolation due to COVID-19 in England: a longitudinal observational study. Lancet Psychiatry. 2021 Feb;8(2):141-149. doi: 10.1016/S2215-0366(20)30482-X. Epub 2020 Dec 9. PMID 33308420

DOCUMENTS (1):
  • Informed Consent Form (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT06020170/ICF_000.pdf